CLINICAL TRIAL: NCT07165496
Title: Cell Phones for Bringing Gay Men From Internet to the Health Center
Brief Title: Text Messaging to Promote HIV Testing in Gay Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Principal Investigator, Luis Menacho Alvirio, Principal Investigator, Universidad Peruana Cayetano Heredia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 62406; S6 0541-01-10 (Other Grant/Funding Number: Grand Challenges Canada)
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: HIV Testing
Keywords: HIV testing; HIV prevention; text messaging; men who have sex with men; health information technologies
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Participants received weekly text messages to promote health and HIV testing and were followed and supported by trained healthcare counselors through two-way communication. Participants were able to set up an appointment for HIV testing at no charge.
  Interventions: Behavioral: Text message-based intervention
- Control arm (No Intervention): Participants were able to set up an appointment for HIV testing at no charge.

INTERVENTIONS:
Behavioral: Text message-based intervention — Participants received weekly text messages to promote health and HIV testing and were followed and supported by trained healthcare counselors through two-way communication over a 12-week period. They were able to schedule a free HIV testing appointment at any time up to six months after enrollment.
  Arms: Intervention arm

SUMMARY:
The rate of HIV and other sexually transmitted infections (STIs) remains high among Peruvian men who have sex with men (MSM), and new prevention programs should be developed to reach and provide sexual health services to more MSM. The Internet is a feasible medium both for recruiting participants and for implementing projects with MSM in Lima, Peru. Likewise, in Peru, mobile phones are promising tools for carrying out HIV-related interventions due to the high rate of mobile phone penetration. The Internet is a way to reach MSM who do not attend traditional health centers due to the stigma associated with being homosexual. Since mobile phones can be used to promote health, the investigators proposed to design, implement, and evaluate an intervention using text messages to promote HIV testing among Peruvian MSM recruited online. To achieve this objective, the investigators conducted a randomized controlled trial to assess the efficacy of a text message-based intervention to promote HIV testing among MSM in Lima recruited via the Internet.

ELIGIBILITY:
Inclusion Criteria:

* Be male at birth
* Be 18 years of age or older
* Be a resident of Lima, Peru
* Report having had sex (oral or anal) with another man in the past 12 months
* Provide informed consent
* Own a mobile phone

Exclusion Criteria:

* Report being HIV-positive
* Have taken an HIV test within the past year

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants who received an HIV test | From enrollment to the end of the 6-month follow-up period
  Having undergone HIV testing at one of the study-affiliated health centers

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Peruana Cayetano Heredia, Lima, Lima Province, Peru

IPD SHARING:
Plan to Share IPD: No